CLINICAL TRIAL: NCT06438458
Title: Effect of Postural Change on Hemoglobin Level in Patients on the Intensive Care Unit
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deventer Ziekenhuis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: NL86966
Record Dates: First submitted 2024-05-21; First posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Anemia
Keywords: Blood composition; Circulatory physiology
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Intervention Model Description: Blood samples are taken before and after the interventions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hb in different positions (Experimental): Hemoglobin concentration after sitting in bed (passively) for >30 min, and after mobilization to a chair for >30 min
  Interventions: Procedure: Postural change from supine to sitting; Procedure: Mobilization to a chair

INTERVENTIONS:
Procedure: Postural change from supine to sitting — Patients go from supine to sitting position in bed (passive)
Procedure: Mobilization to a chair — Patients go from the bed to sitting in a chair (active)

SUMMARY:
Monitoring hemoglobin levels (Hb) is important to identify anemia in hospitalized patients. Changes in posture and mobilization efforts, as demonstrated by previous research, can lead to significant shifts in Hb concentrations. This phenomenon has not been studied in ICU patients.

This study aims to investigate whether postural changes and mobilisation affect Hb in ICU patients. We hypothesize that significant Hb shifts may occur, potentially leading to misinterpretations of anemia and unnecessary diagnostic and therapeutic workup. Understanding this impact can guide clinical practice and prevent unwarranted interventions.

DETAILED DESCRIPTION:
Rationale:

Monitoring hemoglobin levels (Hb) is important to identify anemia in hospitalized patients. Changes in posture and mobilization efforts, as demonstrated by previous research, can lead to significant shifts in Hb concentrations. Low Hb levels due to these shifts are termed 'postural pseudoanemia'.

This phenomenon has not been studied in ICU patients. Many factors may affect Hb concentrations in ICU patients, including plasma volume shifts, bleeding, repeated phlebotomies, hemolysis, bone marrow suppression and functional iron deficiency. When this leads to significant anemia, patients may be treated with red blood cell transfusions. However, blood transfusions have been associated with adverse reactions and should only be performed for appropriate indications. If postural pseudoanemia occurs in ICU patients this could lead to patient harm through inadvertent investigations and red blood cell transfusions. The occurrence of postural pseudoanemia in ICU patients may differ from previous studies because ICU patients are more frequently immobilized for more prolonged periods.

This study aims to investigate whether postural changes affect Hb in ICU patients. We hypothesize that significant Hb shifts may occur, potentially leading to misinterpretations of anemia and unnecessary diagnostic and therapeutic workup. Understanding this impact can guide clinical practice and prevent unwarranted interventions.

Objective:

Main objective: To assess Hb levels in ICU patients upon a change in posture from supine to upright and following mobilization to a chair.

Secondary objectives:

To seek correlations between hemoglobin shifts and changes in serum albumin concentrations upon a change in posture from supine to sitting and following mobilization to a chair.

To seek correlations between hemoglobin shifts and changes in serum uric acid concentrations upon a change in posture from supine to sitting and following mobilization to a chair.

To seek correlations between hemoglobin shifts and levels of CRP and ESR upon a change in posture from supine to sitting and following mobilization to a chair.

To compare hemoglobin concentrations following > 6 hours in supine position at 24 hours with pre-intervention levels for patients remaining in the ICU.

Any other changes seen in the lab measurements or vital parameters upon a change in posture?

Study design:

Prospective uncontrolled interventional study.

Study population:

Patients > 18 years old, admitted to the intensive care unit.

Intervention:

All patients will undergo a change in posture from supine to upright, followed by mobilization to a chair.

Main study parameters/endpoints:

Relative percentage change in Hb.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years, of any gender and ethnic background
* Admitted to the intensive care unit
* Able to give informed consent
* Patients with an arterial line as part of their treatment plan.
* Patients able to remain seated in chair for at least 30 minutes
* Patients able to remain supine overnight for at least 6 hours

Exclusion Criteria:

* Delirium or inability to give informed consent
* Inability to understand written information in Dutch
* Patients on artificial ventilation
* Orotracheally intubated patients (spontaneous breathing through a tracheostomy cannula is allowed)
* Patients treated with noradrenaline > 0.05 ug/kg/min
* Patients treated with argipressin
* Patients who received a blood transfusion within 24 hours before measurements
* Patients who received > 3 L of fluids within 24 hours before measurements
* Patients who received > 500 ml of iv fluids within 4 hours of measurements
* Severe restlessness or inability to remain supine for 6 hours before initial blood sampling
* Patients being treated with diuretics
* Patients admitted with:
* Decompensated right heart failure
* Pulmonary hypertension
* Pulmonary embolism
* Active bleeding or risk of >100 ml blood loss
* Hematological disorder/malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin | 3 hours
  Hemoglobin concentration

SECONDARY OUTCOMES:
Albumin | 3 hours
  Albumin concentration

OTHER OUTCOMES:
Uric acid | 3 hours
  Uric acid concentration

CONTACTS AND LOCATIONS:
Overall Officials: Alfred L van Steveninck, M.D., Ph.D., Principal Investigator — Deventer Ziekenhuis
Locations (1):
- Deventer Hospital, Deventer, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data can be obtained from the principal investigator upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After preparation of the manuscript.
Access Criteria: A written request must be sent to the principal investigator.